CLINICAL TRIAL: NCT06625879
Title: Efficacy of the Mid-point Transverse Process to Pleura Block Versus Serratus Anterior Plane Block for Postoperative Analgesia After Modified Radical Mastectomy as a Randomized Trial
Brief Title: The Mid-point Transverse Process to Pleura Block Versus Serratus Anterior Plane Block for Postoperative Analgesia After Modified Radical Mastectomy
Acronym: (SAPB) (MTPB)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alaa Ashraf Hassan Abd Elsalam, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD325/2023
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: (Serratus Anterior Plane Block (SAPB) Group) (n=15) (Active Comparator): Group I: (Serratus Anterior Plane Block (SAPB) Group) (n=15):
  The patient will lay on her side with arm brought forward, the linear US transducer probe (10-12 MHz) will be placed in the midaxillary line and then moved caudal from second rib until the sixth intercostal space. At this point, the subcutaneous tissue and serratus muscle will be identified in the superficial plane, whereas the external intercostal muscles will be identified in the intermediate plane and finally in the deep plane the ribs, pleura and lung will be identified. The needle will be advanced from caudal to cranial direction. In-plane technique will be used until the tip of the needle placed between the serratus anterior muscle and the external intercostal muscle (deep SABP) (Blanco et al., 2013). A volume of titrated bolus of 20 ml of bupivacaine 0.5% will be injected after aspiration to avoid intravascular injection (Lin J et al., 2020).
  Interventions: Procedure: Serratus Anterior Plane Block (SAPB)
- GroupII: (Midpoint transverse process to pleura (MTP) block group )(n=15) (Active Comparator): GroupII: (Midpoint transverse process to pleura (MTP) block group )(n=15):
  In the lateral postion, the T4 spine will be counted by ultrasound, and high frequency linear US transducer probe (10-12 MHz) will be placed longitudinally, approximately 2.5 cm lateral to the midline the needle will be advanced in plane from cranial to caudal direction. The desired end point for the needle tip will be the midpoint of the line between the posterior border of the transverse process of T4 and the pleura(injection will be deep (anterior) to the posterior aspect of the vertebral transverse process but superficial to the superior costotransverse ligment),the needle tip dose not enter the paravertebral space (Chin et al., 2021), a volume of titrated bolus of 20 ml of bupivacaine 0.5% will be injected after aspiration to avoid intravascular injection,pleural displacement and bowing of erector spinae will be observed at the side of injection (Syal et al., 2020; Pusch et al., 2000).
  Interventions: Procedure: Midpoint transverse process to pleura (MTP) block

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block (SAPB) — Group I: (Serratus Anterior Plane Block (SAPB) Group) (n=15):
  The patient will lay on her side with arm brought forward, the linear US transducer probe (10-12 MHz) will be placed in the midaxillary line and then moved caudal from second rib until the sixth intercostal space. At this point, the subcutaneous tissue and serratus muscle will be identified in the superficial plane, whereas the external intercostal muscles will be identified in the intermediate plane and finally in the deep plane the ribs, pleura and lung will be identified. The needle will be advanced from caudal to cranial direction. In-plane technique will be used until the tip of the needle placed between the serratus anterior muscle and the external intercostal muscle (deep SABP) . A volume of titrated bolus of 20 ml of bupivacaine 0.5% will be injected after aspiration to avoid intravascular injection.
  Arms: Group I: (Serratus Anterior Plane Block (SAPB) Group) (n=15)
Procedure: Midpoint transverse process to pleura (MTP) block — In the lateral postion, the T4 spine will be counted by ultrasound, and high frequency linear US transducer probe (10-12 MHz) will be placed longitudinally, approximately 2.5 cm lateral to the midline the needle will be advanced in plane from cranial to caudal direction. The desired end point for the needle tip will be the midpoint of the line between the posterior border of the transverse process of T4 and the pleura(injection will be deep (anterior) to the posterior aspect of the vertebral transverse process but superficial to the superior costotransverse ligment),the needle tip dose not enter the paravertebral space , a volume of titrated bolus of 20 ml of bupivacaine 0.5% will be injected after aspiration to avoid intravascular injection,pleural displacement and bowing of erector spinae will be observed at the side of injection .
  Arms: GroupII: (Midpoint transverse process to pleura (MTP) block group )(n=15)

SUMMARY:
Several studies proved that the serratus anterior plane block(SAPB) offer analgesia not inferior or as effective to opioids which is mainstay of analgesia (chai et al., 2023).

In this study we will compare the analgesic effect of the serratus anterior plane block versus a new paraspinal technique block which is the midpoint transverse process to pleura (MTP) block for postoperative analgesia after modefied radical mastectomy.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women both in the developed and less developed world. In 2012, it represented about 12 percent of all new cancer cases and 25 percent of all cancers in women (Jain et al., 2020).

Surgery is one of the mainstays of treatment, and a procedure called modified radical mastectomy (MRM) is now a standard surgical treatment for early stage breast cancers.These procedures cause significant acute pain and may progress to chronic pain states in 25-60% of cases (Andersen and Kehlet, 2011).

Though various risk factors have been suggested, inappropriate acute postoperative pain management has been associated with the development of chronic post mastectomy pain, a complex post-surgical pain syndrome that may occur following any type of breast surgery (Macrea, 2001). The traditional opioid based analgesia remains the mainstay, however. Different techniques including regional local anaesthetic infiltration, paravertebral and neuroaxial analgesia, anti_neuropathic analgesics and NMDA antagonists have all been used either singly or in combination, (Macrea, 2001). Post operative pain is usually acute nociceptive pain, it occurs as normal response to noxious insult or injury (Dworkin et al., 2007) .

Inadequately controlled pain negatively affects quality of life, functional recovery and increase the risk for post-surgical complications (Apfelbaum, 2003).

After the application of ultrasound in anaesthetic practice,several blocks have been described recently,Serratus anterior plane blocks performed at the axillary fossa within a region bounded by the anterior and posterior axillary lines and th 3rd to 6th ribs (Chin et al., 2021), in which the intercostobrachialis nerve, lateral cutaneous branches of the intercostal nerves (T2-T9),long thoracic nerve,and the thoracodorsal nerve are located in a compartment between the serratus anterior and the latissimus dorsi muscles (Blanco et al., 2013).

The MTP block described by Costache et al. (2017) is a new block described for thoracic surgery, it involves deposition of the local anesthetic drug midway between the transverse process and the pleura. Postulated that the local anesthetic deposited at this point will reach the paravertebral space through several possible mechanisms, such as medially through the gap between the superior costotransverse ligament (SCTL) and vertebral bodies, through fenestrations in SCTL, and laterally through the internal intercostal membrane, the neural target will be the dorsal and ventral rami of spinal nerves, spanning 1-3 levels cranial and caudal to the level of injection,the advantage of the MTP block over the conventional thoracic paravertebral block is that the visualization of SCTL is not required, which might be difficult in patients with obesity. The second advantage is that the target point of the needle is very superficial and far from structures, such as the pleura and neurovascular bundles ,making this novel block much safer (Syal et al., 2020).

2.AIM / OBJECTIVES

The aim of work is to evaluate The Effectiveness of Ultrasound Guided mid-point transverse process to pleura block versus the serratus anterior plane block for postoperative analgesia after modefied radical mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing unilateral Modified Radical Mastectomy. Physical status: ASA grades I and II. Age between 35 and 60 years old.

Exclusion Criteria:

* Known Allergy to one of the study drugs. Asthmatic patients. Patients undergoing bilateral Modified Radical Mastectomy. Patients refusal of procedure or participation in the study. ASA classes III or above. Local skin infection at the site of the block. Pregnant Patients. Other malignancy. History or evidence of coagulopathy. History of use of anti coagulant or anti platelet therapy. Body mass index ≥40 kg/m2.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients will undergoing modefied radical mastectomy
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
the mean duration to require first rescue analgesia which will be (Diclofenac 75mg) when NRS pain score ≥4 at rest. | 24 hours post- operative
  the mean duration to require first rescue analgesia which will be (Diclofenac 75mg) when NRS pain score ≥4 at rest. If no response within 1 hour pethidine 50mg IM will be given. If NRS pain score is ≥4 at rest after 2 hours another dose of pethidine 25mg IM will be given.

SECONDARY OUTCOMES:
The total number of doses of the rescue analgesia that will be received in the 24 hours postoperatively if the NRS pain score at rest ≥4 | 24 hours post- operative
  The total number of doses of the rescue analgesia that will be received in the 24 hours postoperatively if the NRS pain score at rest ≥4, NRS at rest and at movement (cough or rotating the body), a 4-point objective pain score (OPS),hemodynamics and side effects (nausea and vomiting)